CLINICAL TRIAL: NCT03636945
Title: Evaluation of the Clinical Performance of 18F-FDOPA PET-CT in the Preoperative Initial Assessment of Medullary Thyroid Carcinoma: Multicenter Prospective Study
Brief Title: Evaluation of 18F-FDOPA PET-CT in the Preoperative Initial Assessment of Medullary Thyroid Carcinoma
Acronym: TEPCMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-10
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Medullary Thyroid Carcinoma
MeSH Terms: conditions — Carcinoma, Medullary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medullary thyroid carcinoma (Experimental): Patients with MTC who have serum calcitonin> 150 pg / ml at initial diagnosis and have performed baseline imaging examinations within the last 3 months will be included in the study A PET at 18F-FDOPA will be performed according to a very powerful acquisition protocol
  Interventions: Other: PET at 18F-FDOPA

INTERVENTIONS:
Other: PET at 18F-FDOPA — 18F-fluorodihydroxyphenylalanine (18F-FDOPA) PET imaging

SUMMARY:
Medullary thyroid carcinoma (MTC) develops at the expense of calcitonin cells and is often characterized by lymph node metastases and sometimes visceral metastases. Improvement of preoperative diagnosis is of major importance in CMT because the quality of the initial surgery determines the prognosis. In recent years, 18F-fluorodihydroxyphenylalanine (18F-FDOPA) PET / CT was considered the most sensitive functional imaging tool in the evaluation of persistent CMT. To date, 18F-FDOPA PET at initial diagnosis has been reported in a few clinical cases.

The main objective is to demonstrate that 18F-FDOPA PET provides additional information compared to conventional imaging on the initial diagnosis of CMT patients.

The secondary objectives are to describe the nature of the information provided by PET / CT imaging, the main factors influencing tracer uptake and the positivity of PET / CT, and the impact of the examination on the care of the patient.

This is a prospective, multicenter and open study.

Patients with TCM who have serum calcitonin> 150 pg / ml at initial diagnosis and have performed baseline imaging examinations within the last 3 months will be included in the study . A PET at 18F-FDOPA will be performed according to a very powerful acquisition protocol. Image analysis will be performed blindly from the results of conventional imaging. All exams will be compared, in accordance with the gold standard. Therapeutic intentions will be collected before and after the PET imaging, as well as the actual management in place.

DETAILED DESCRIPTION:
Medullary thyroid carcinoma (MTC) develops at the expense of calcitonin cells and is often characterized by lymph node metastases (> 50% of cases) and sometimes visceral metastases (> 5%). Improvement of preoperative diagnosis is of major importance in CMT because the quality of the initial surgery determines the prognosis. In recent years, 18F-fluorodihydroxyphenylalanine (18F-FDOPA) PET / CT was considered the most sensitive functional imaging tool in the evaluation of persistent CMT. To date, 18F-FDOPA PET at initial diagnosis has been reported in a few clinical cases. Preliminary study, which included 9 CMT patients, 18F-FDOPA PET showed very promising results during the initial diagnosis, particularly in node staging.

The main objective is to demonstrate that 18F-FDOPA PET provides additional information compared to conventional imaging on the initial diagnosis of CMT patients. The secondary objectives are to describe the nature of the information provided by PET / CT imaging, the main factors influencing tracer uptake and the positivity of PET / CT, and the impact of the examination on the care of the patient.

This is a prospective, multicenter and open study.

Patients with TCM who have serum calcitonin> 150 pg / ml at initial diagnosis and have performed baseline imaging examinations (as recommended by the 2015 ATA) within the last 3 months will be included in the study . A PET at 18F-FDOPA will be performed according to a very powerful acquisition protocol. Image analysis will be performed blindly from the results of conventional imaging. All exams will be compared, in accordance with the gold standard. Therapeutic intentions will be collected before and after the PET imaging, as well as the actual management in place.

Number of patients expected: 62. Duration of the study: 29 months of inclusion and 7 months of follow-up.

About 60 to 70 patients with a CMT are operated annually in the centers involved. Nuclear physicians, endocrine surgeons, endocrinologists and anatomopathologists work together in institutional and interinstitutional team meetings (SFE-RENATEN). Some of the centers have already collaborated on the implementation of a large PHRC-INCa project recently published in the JCEM.

ELIGIBILITY:
Inclusion Criteria:

* Major patient, affiliated to a social security scheme and having signed a written consent
* Patients with CMT (initial diagnosis)
* Serum calcitonin> 150 μg / ml
* Patient who had the baseline imaging assessment during the 3 months preceding the 18F-FDOPA PET scan (as recommended by the 2015 ATA (11)), according to the serum calcitonin level:

  * 150 <Calcitonin <500: cervical ultrasound + cervico-thoracic CT scan
  * Calcitonin ≥500: cervical ultrasound, cervico-thoracoabdominopelvic CT scan, bone MRI.

Exclusion Criteria:

* Pregnant women (positive pregnancy test) or lactating women can not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
number of patient with aditionnal information | 90 MINUTES
  the proportion of CMT patients for whom 18F-FDOPA PET / CT PET provides additional information compared to the conventional imaging (CI) assessment at the initial diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France